CLINICAL TRIAL: NCT02363647
Title: Personalized Cancer Therapy for Patients With Metastatic Medullary Thyroid or Metastatic Colon Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: No Current Funding
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Krzysztof Misiukiewicz, Assistant Professor, Medicine, Hematology and Medical Oncology, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO#1: 15-0146
Record Dates: First submitted 2015-02-03; First posted 2015-02-16 (Estimated); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Medullary Thyroid Cancer; Colon Cancer
Keywords: medullary thyroid cancer; thyroid cancer; personalized therapy; personalized chemotherapy; individualized treatment; colon cancer; colorectal cancer
MeSH Terms: conditions — Carcinoma, Medullary; Colonic Neoplasms; Thyroid Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tumor Genomic Analysis (Experimental): Personalized Therapy Plan Patients with Metastatic Medullary or Colon Cancer being treated with the Personalized Treatment Plan developed during the different tumor genomic analysis study.
  Interventions: Other: Tumor Genomic Analysis

INTERVENTIONS:
Other: Tumor Genomic Analysis — Tumor mutations identified by deep DNA and RNA sequencing of individual tumors are screened for tumor drivers, which are then incorporated into the "personal" Drosophila model and tested against a library of FDA approved drugs. Fly mortality is used as a surrogate for toxicity and increased survival to adulthood; improvements in tumor mutation-linked eye and/or wing abnormalities serve to quantify efficacy. This allows rapid and parallel screening of FDA approved drugs and subsequent drug combinations. The most efficacious and least toxic combinations are tested in xenograft models and a multidisciplinary tumor board of experts select the best therapeutic option. The objective is to demonstrate that the personalized drosophila model approach is superior to the current standard. Patient will be offered an unique "personalized" single drug or combination of drugs, all FDA approved, based on the Drosophila drug screening process.

SUMMARY:
The Personalized Discovery Process is the only program offering patients treatment recommendations based on an empirically constructed Drosophila "fly" model of their disease. Special committee selects one of the one of the few 2-3 FDA approved drug combinations or single agents that improved survival in the fly cancer model.

DETAILED DESCRIPTION:
Tumor mutations identified by deep DNA and RNA sequencing of individual tumors are screened for tumor drivers, which are then incorporated into the "personal" Drosophila model and tested against a library of FDA approved drugs. Fly mortality is used as a surrogate for toxicity and increased survival to adulthood; improvements in tumor mutation-linked eye and/or wing abnormalities serve to quantify efficacy. This allows rapid and parallel screening of FDA approved drugs and subsequent drug combinations. The most efficacious and least toxic combinations are tested in xenograft models and a multidisciplinary tumor board of experts select the best therapeutic option. The objective is to demonstrate that the personalized drosophila model approach is superior to the current standard used in medullary thyroid or colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients already enrolled to the separate Tumor Genomic Analysis and Molecular Testing for Personalized Cancer Therapy study, for which a personalized therapeutic plan has been successfully created under that protocol and selected by the multidisciplinary tumor board of experts for use in this therapeutic clinical trial
* Histologically confirmed MTC by a Mount Sinai pathologist
* Recurrent/metastatic or incurable MTC
* Age > 18 years old
* Life expectancy must exceed 1 year from enrollment in the study
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≤ 2
* The subject has documented worsening of disease (progressive disease) at screening compared with a previous CT scan or MRI image done within 14 months of screening Documentation of progression may be made by CT, MRI, or PET assessment
* Adequate organ and bone marrow function defined by routine testing
* The subject has no other diagnosis of cancer (unless non-melanoma skin cancer, an early form of cervical cancer, or another cancer diagnosed ≥ 2 years previously) and currently has no evidence of active other malignancy (unless non-melanoma skin cancer or an early form of cervical cancer)
* Signed and dated informed consent form indicating that the patient has been informed of all pertinent aspects of the trial prior to enrolment

Exclusion Criteria:

* Patients who are currently receiving and responding to a different course of anti-neoplastic therapy, within the limits of acceptable toxicity per standard clinical practice, may not be enrolled to this study
* Current symptomatic brain metastases. If previously present, the metastases must have been treated at least two months before participation in this study. CT or MRI scan of the brain is mandatory to assess the presence or not of brain metastases
* History of other malignancy within the last 5 years, except for adequately treated carcinoma in situ of the cervix or basal cell, or squamous cell carcinoma of the skin
* History of significant cardiac disease defined as:

  * Symptomatic CHF (NYHA classes III-IV)
  * High-risk uncontrolled arrhythmias; i.e. atrial tachycardia with a heart rate > 100/min at rest, significant ventricular arrhythmia or higher-grade AV-block (second degree AV-block Type 2 [Mobitz 2] or third degree AV-block)
  * Prolongation of QT interval > 480 msecs
  * History of myocardial infarction within last 12 months
  * Clinically significant valvular heart disease
  * Angina pectoris requiring anti-angina treatment
  * Current uncontrolled hypertension (persistent systolic > 180 mmHg and/or diastolic > 100 mmHg). Initiation or adjustment of antihypertensive medication is permitted prior to study entry
* Evidence of active bleeding or bleeding diathesis
* Cerebrovascular accident at any time in the past, transient ischemic attack, deep venous thrombosis or pulmonary embolism in the past 6 months
* Current severe, uncontrolled systemic disease
* Presence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule
* Failure to use contraception in patients with preserved reproductive capacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-01; Primary Completion 2022-08 (Actual); Study Completion 2022-08 (Actual)

PRIMARY OUTCOMES:
Overall response rate (ORR) | up to 3 years
  ORR as the sum of partial responses (PRs) and complete responses (CRs)

SECONDARY OUTCOMES:
Progression-free Survival (PFS) | up to 3 years
  The length of time during and after the treatment of disease that a patient lives with the disease but it does not get worse.
Overall survival (OS) | up to 3 years
  The length of time from either the date of diagnosis or the start of treatment for disease, that patients diagnosed with the disease are still alive.

CONTACTS AND LOCATIONS:
Overall Officials: Krzysztof Misiukiewicz, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

REFERENCES:
- [Background] Hundahl SA, Fleming ID, Fremgen AM, Menck HR. A National Cancer Data Base report on 53,856 cases of thyroid carcinoma treated in the U.S., 1985-1995 [see commetns]. Cancer. 1998 Dec 15;83(12):2638-48. doi: 10.1002/(sici)1097-0142(19981215)83:123.0.co;2-1. PMID 9874472
- [Background] Saad MF, Ordonez NG, Rashid RK, Guido JJ, Hill CS Jr, Hickey RC, Samaan NA. Medullary carcinoma of the thyroid. A study of the clinical features and prognostic factors in 161 patients. Medicine (Baltimore). 1984 Nov;63(6):319-42. PMID 6503683
- [Background] Zedenius J, Larsson C, Bergholm U, Bovee J, Svensson A, Hallengren B, Grimelius L, Backdahl M, Weber G, Wallin G. Mutations of codon 918 in the RET proto-oncogene correlate to poor prognosis in sporadic medullary thyroid carcinomas. J Clin Endocrinol Metab. 1995 Oct;80(10):3088-90. doi: 10.1210/jcem.80.10.7559902.
- [Background] Elisei R, Cosci B, Romei C, Bottici V, Renzini G, Molinaro E, Agate L, Vivaldi A, Faviana P, Basolo F, Miccoli P, Berti P, Pacini F, Pinchera A. Prognostic significance of somatic RET oncogene mutations in sporadic medullary thyroid cancer: a 10-year follow-up study. J Clin Endocrinol Metab. 2008 Mar;93(3):682-7. doi: 10.1210/jc.2007-1714. Epub 2007 Dec 11. PMID 18073307
- [Background] Romei C, Elisei R, Pinchera A, Ceccherini I, Molinaro E, Mancusi F, Martino E, Romeo G, Pacini F. Somatic mutations of the ret protooncogene in sporadic medullary thyroid carcinoma are not restricted to exon 16 and are associated with tumor recurrence. J Clin Endocrinol Metab. 1996 Apr;81(4):1619-22. doi: 10.1210/jcem.81.4.8636377.
- [Background] Eng C, Clayton D, Schuffenecker I, Lenoir G, Cote G, Gagel RF, van Amstel HK, Lips CJ, Nishisho I, Takai SI, Marsh DJ, Robinson BG, Frank-Raue K, Raue F, Xue F, Noll WW, Romei C, Pacini F, Fink M, Niederle B, Zedenius J, Nordenskjold M, Komminoth P, Hendy GN, Mulligan LM, et al. The relationship between specific RET proto-oncogene mutations and disease phenotype in multiple endocrine neoplasia type 2. International RET mutation consortium analysis. JAMA. 1996 Nov 20;276(19):1575-9. PMID 8918855
- [Background] Ceolin L, Siqueira DR, Romitti M, Ferreira CV, Maia AL. Molecular basis of medullary thyroid carcinoma: the role of RET polymorphisms. Int J Mol Sci. 2012;13(1):221-39. doi: 10.3390/ijms13010221. Epub 2011 Dec 27. PMID 22312249
- [Background] Catalano MG, Fortunati N, Boccuzzi G. Epigenetics modifications and therapeutic prospects in human thyroid cancer. Front Endocrinol (Lausanne). 2012 Mar 19;3:40. doi: 10.3389/fendo.2012.00040. eCollection 2012. PMID 22649419
- [Background] Borrello MG, Ardini E, Locati LD, Greco A, Licitra L, Pierotti MA. RET inhibition: implications in cancer therapy. Expert Opin Ther Targets. 2013 Apr;17(4):403-19. doi: 10.1517/14728222.2013.758715. Epub 2013 Mar 6. PMID 23461584
- [Background] Schlumberger MJ, Elisei R, Bastholt L, Wirth LJ, Martins RG, Locati LD, Jarzab B, Pacini F, Daumerie C, Droz JP, Eschenberg MJ, Sun YN, Juan T, Stepan DE, Sherman SI. Phase II study of safety and efficacy of motesanib in patients with progressive or symptomatic, advanced or metastatic medullary thyroid cancer. J Clin Oncol. 2009 Aug 10;27(23):3794-801. doi: 10.1200/JCO.2008.18.7815. Epub 2009 Jun 29. PMID 19564535
- [Background] Sherman SI. Advances in chemotherapy of differentiated epithelial and medullary thyroid cancers. J Clin Endocrinol Metab. 2009 May;94(5):1493-9. doi: 10.1210/jc.2008-0923. Epub 2009 Mar 3. PMID 19258410
- [Background] Bible KC, Suman VJ, Molina JR, Smallridge RC, Maples WJ, Menefee ME, Rubin J, Sideras K, Morris JC 3rd, McIver B, Burton JK, Webster KP, Bieber C, Traynor AM, Flynn PJ, Goh BC, Tang H, Ivy SP, Erlichman C; Endocrine Malignancies Disease Oriented Group; Mayo Clinic Cancer Center; Mayo Phase 2 Consortium. Efficacy of pazopanib in progressive, radioiodine-refractory, metastatic differentiated thyroid cancers: results of a phase 2 consortium study. Lancet Oncol. 2010 Oct;11(10):962-72. doi: 10.1016/S1470-2045(10)70203-5. Epub 2010 Sep 17. PMID 20851682
- [Background] Wells SA Jr, Robinson BG, Gagel RF, Dralle H, Fagin JA, Santoro M, Baudin E, Elisei R, Jarzab B, Vasselli JR, Read J, Langmuir P, Ryan AJ, Schlumberger MJ. Vandetanib in patients with locally advanced or metastatic medullary thyroid cancer: a randomized, double-blind phase III trial. J Clin Oncol. 2012 Jan 10;30(2):134-41. doi: 10.1200/JCO.2011.35.5040. Epub 2011 Oct 24. PMID 22025146
- [Background] Schoffski P, E.R., Muller S, Brose MS, Shah MH, Licitra LF, An international, double-blind, randomized, placebo-controlled phase III trial (EXAM) of cabozantinib (XL184) in medullary thyroid carcinoma (MTC) patients with documented RECIST progression at baseline. ASCO 2012, June 1-5, 2012.
- [Background] Read RD, Goodfellow PJ, Mardis ER, Novak N, Armstrong JR, Cagan RL. A Drosophila model of multiple endocrine neoplasia type 2. Genetics. 2005 Nov;171(3):1057-81. doi: 10.1534/genetics.104.038018. Epub 2005 Jun 18. PMID 15965261
- [Background] Kjaer S, Kurokawa K, Perrinjaquet M, Abrescia C, Ibanez CF. Self-association of the transmembrane domain of RET underlies oncogenic activation by MEN2A mutations. Oncogene. 2006 Nov 9;25(53):7086-95. doi: 10.1038/sj.onc.1209698. Epub 2006 May 29. PMID 16732321
- [Background] Cakir M, Grossman AB. Medullary thyroid cancer: molecular biology and novel molecular therapies. Neuroendocrinology. 2009;90(4):323-48. doi: 10.1159/000220827. Epub 2009 May 25. PMID 19468197
- [Background] Segouffin-Cariou C, Billaud M. Transforming ability of MEN2A-RET requires activation of the phosphatidylinositol 3-kinase/AKT signaling pathway. J Biol Chem. 2000 Feb 4;275(5):3568-76. doi: 10.1074/jbc.275.5.3568. PMID 10652352
- [Background] Das T, Cagan R. Drosophila as a novel therapeutic discovery tool for thyroid cancer. Thyroid. 2010 Jul;20(7):689-95. doi: 10.1089/thy.2010.1637. PMID 20578898
- [Background] Vidal M, Larson DE, Cagan RL. Csk-deficient boundary cells are eliminated from normal Drosophila epithelia by exclusion, migration, and apoptosis. Dev Cell. 2006 Jan;10(1):33-44. doi: 10.1016/j.devcel.2005.11.007. PMID 16399076
- [Background] Wells SA Jr, Gosnell JE, Gagel RF, Moley J, Pfister D, Sosa JA, Skinner M, Krebs A, Vasselli J, Schlumberger M. Vandetanib for the treatment of patients with locally advanced or metastatic hereditary medullary thyroid cancer. J Clin Oncol. 2010 Feb 10;28(5):767-72. doi: 10.1200/JCO.2009.23.6604. Epub 2010 Jan 11. PMID 20065189
- [Background] Vidal M, Wells S, Ryan A, Cagan R. ZD6474 suppresses oncogenic RET isoforms in a Drosophila model for type 2 multiple endocrine neoplasia syndromes and papillary thyroid carcinoma. Cancer Res. 2005 May 1;65(9):3538-41. doi: 10.1158/0008-5472.CAN-04-4561. PMID 15867345
- [Background] Haura EB, Ricart AD, Larson TG, Stella PJ, Bazhenova L, Miller VA, Cohen RB, Eisenberg PD, Selaru P, Wilner KD, Gadgeel SM. A phase II study of PD-0325901, an oral MEK inhibitor, in previously treated patients with advanced non-small cell lung cancer. Clin Cancer Res. 2010 Apr 15;16(8):2450-7. doi: 10.1158/1078-0432.CCR-09-1920. Epub 2010 Mar 23. PMID 20332327
- [Background] O'Brien SG, Guilhot F, Larson RA, Gathmann I, Baccarani M, Cervantes F, Cornelissen JJ, Fischer T, Hochhaus A, Hughes T, Lechner K, Nielsen JL, Rousselot P, Reiffers J, Saglio G, Shepherd J, Simonsson B, Gratwohl A, Goldman JM, Kantarjian H, Taylor K, Verhoef G, Bolton AE, Capdeville R, Druker BJ; IRIS Investigators. Imatinib compared with interferon and low-dose cytarabine for newly diagnosed chronic-phase chronic myeloid leukemia. N Engl J Med. 2003 Mar 13;348(11):994-1004. doi: 10.1056/NEJMoa022457. PMID 12637609
- [Background] Boss DS, Beijnen JH, Schellens JH. Clinical experience with aurora kinase inhibitors: a review. Oncologist. 2009 Aug;14(8):780-93. doi: 10.1634/theoncologist.2009-0019. Epub 2009 Aug 14. PMID 19684075
- [Background] Kantarjian H, Talpaz M, O'Brien S, Garcia-Manero G, Verstovsek S, Giles F, Rios MB, Shan J, Letvak L, Thomas D, Faderl S, Ferrajoli A, Cortes J. High-dose imatinib mesylate therapy in newly diagnosed Philadelphia chromosome-positive chronic phase chronic myeloid leukemia. Blood. 2004 Apr 15;103(8):2873-8. doi: 10.1182/blood-2003-11-3800. Epub 2003 Dec 24. PMID 15070658
- [Background] Knight ZA, Lin H, Shokat KM. Targeting the cancer kinome through polypharmacology. Nat Rev Cancer. 2010 Feb;10(2):130-7. doi: 10.1038/nrc2787. PMID 20094047
- [Background] Karaman MW, Herrgard S, Treiber DK, Gallant P, Atteridge CE, Campbell BT, Chan KW, Ciceri P, Davis MI, Edeen PT, Faraoni R, Floyd M, Hunt JP, Lockhart DJ, Milanov ZV, Morrison MJ, Pallares G, Patel HK, Pritchard S, Wodicka LM, Zarrinkar PP. A quantitative analysis of kinase inhibitor selectivity. Nat Biotechnol. 2008 Jan;26(1):127-32. doi: 10.1038/nbt1358. PMID 18183025
- [Background] Wilhelm S, Carter C, Lynch M, Lowinger T, Dumas J, Smith RA, Schwartz B, Simantov R, Kelley S. Discovery and development of sorafenib: a multikinase inhibitor for treating cancer. Nat Rev Drug Discov. 2006 Oct;5(10):835-44. doi: 10.1038/nrd2130. PMID 17016424
- [Background] Hirabayashi S, Baranski TJ, Cagan RL. Transformed Drosophila cells evade diet-mediated insulin resistance through wingless signaling. Cell. 2013 Aug 1;154(3):664-75. doi: 10.1016/j.cell.2013.06.030. PMID 23911328
- [Background] Dar AC, Das TK, Shokat KM, Cagan RL. Chemical genetic discovery of targets and anti-targets for cancer polypharmacology. Nature. 2012 Jun 6;486(7401):80-4. doi: 10.1038/nature11127. PMID 22678283
- [Background] Markstein M, Dettorre S, Cho J, Neumuller RA, Craig-Muller S, Perrimon N. Systematic screen of chemotherapeutics in Drosophila stem cell tumors. Proc Natl Acad Sci U S A. 2014 Mar 25;111(12):4530-5. doi: 10.1073/pnas.1401160111. Epub 2014 Mar 10. PMID 24616500
- [Background] Karp JE, Thomas BM, Greer JM, Sorge C, Gore SD, Pratz KW, Smith BD, Flatten KS, Peterson K, Schneider P, Mackey K, Freshwater T, Levis MJ, McDevitt MA, Carraway HE, Gladstone DE, Showel MM, Loechner S, Parry DA, Horowitz JA, Isaacs R, Kaufmann SH. Phase I and pharmacologic trial of cytosine arabinoside with the selective checkpoint 1 inhibitor Sch 900776 in refractory acute leukemias. Clin Cancer Res. 2012 Dec 15;18(24):6723-31. doi: 10.1158/1078-0432.CCR-12-2442. Epub 2012 Oct 23. PMID 23092873
- [Background] Willoughby LF, Schlosser T, Manning SA, Parisot JP, Street IP, Richardson HE, Humbert PO, Brumby AM. An in vivo large-scale chemical screening platform using Drosophila for anti-cancer drug discovery. Dis Model Mech. 2013 Mar;6(2):521-9. doi: 10.1242/dmm.009985. Epub 2012 Sep 20. PMID 22996645
- [Background] Dancey JE, Chen HX. Strategies for optimizing combinations of molecularly targeted anticancer agents. Nat Rev Drug Discov. 2006 Aug;5(8):649-59. doi: 10.1038/nrd2089. PMID 16883303
- [Background] Tentler JJ, Tan AC, Weekes CD, Jimeno A, Leong S, Pitts TM, Arcaroli JJ, Messersmith WA, Eckhardt SG. Patient-derived tumour xenografts as models for oncology drug development. Nat Rev Clin Oncol. 2012 Apr 17;9(6):338-50. doi: 10.1038/nrclinonc.2012.61. PMID 22508028
- [Background] Tsimberidou AM, Iskander NG, Hong DS, Wheler JJ, Falchook GS, Fu S, Piha-Paul S, Naing A, Janku F, Luthra R, Ye Y, Wen S, Berry D, Kurzrock R. Personalized medicine in a phase I clinical trials program: the MD Anderson Cancer Center initiative. Clin Cancer Res. 2012 Nov 15;18(22):6373-83. doi: 10.1158/1078-0432.CCR-12-1627. Epub 2012 Sep 10. PMID 22966018
- [Background] Wheler JJ, Tsimberidou AM, Hong DS, Naing A, Falchook GS, Fu S, Moulder S, Stephen B, Wen S, Kurzrock R. Risk of serious toxicity in 1181 patients treated in phase I clinical trials of predominantly targeted anticancer drugs: the M. D. Anderson Cancer Center experience. Ann Oncol. 2012 Aug;23(8):1963-1967. doi: 10.1093/annonc/mds027. Epub 2012 Feb 29. PMID 22377564
- [Background] Annas GJ. The changing landscape of human experimentation: Nuremberg, Helsinki, and beyond. Health Matrix Clevel. 1992 Summer;2(2):119-40. No abstract available. PMID 10124876
- [Background] Decoster G, Stein G, Holdener EE. Responses and toxic deaths in phase I clinical trials. Ann Oncol. 1990;1(3):175-81. doi: 10.1093/oxfordjournals.annonc.a057716. PMID 2148104
- [Background] Dehan P, Kustermans G, Guenin S, Horion J, Boniver J, Delvenne P. DNA methylation and cancer diagnosis: new methods and applications. Expert Rev Mol Diagn. 2009 Oct;9(7):651-7. doi: 10.1586/erm.09.53. PMID 19817550
- [Background] Bosserman L, Prendergast F, Herbst R, Fleisher M, Salom E, Strickland S, Raptis A, Hallquist A, Perree M, Rajurkar S, Karimi M, Rogers K, Davidson D, Willis C, Penalver M, Homesley H, Burrell M, Garrett A, Rutledge J, Chernick M, Presant CA. The microculture-kinetic (MiCK) assay: the role of a drug-induced apoptosis assay in drug development and clinical care. Cancer Res. 2012 Aug 15;72(16):3901-5. doi: 10.1158/0008-5472.CAN-12-0681. Epub 2012 Aug 3. PMID 22865459
- [Background] Arrowsmith J. Trial watch: Phase II failures: 2008-2010. Nat Rev Drug Discov. 2011 May;10(5):328-9. doi: 10.1038/nrd3439. No abstract available. PMID 21532551
- [Background] Arrowsmith J. Trial watch: phase III and submission failures: 2007-2010. Nat Rev Drug Discov. 2011 Feb;10(2):87. doi: 10.1038/nrd3375. No abstract available. PMID 21283095
- [Background] Evans WE, Relling MV. Pharmacogenomics: translating functional genomics into rational therapeutics. Science. 1999 Oct 15;286(5439):487-91. doi: 10.1126/science.286.5439.487. PMID 10521338
- [Background] Joensuu H, Roberts PJ, Sarlomo-Rikala M, Andersson LC, Tervahartiala P, Tuveson D, Silberman S, Capdeville R, Dimitrijevic S, Druker B, Demetri GD. Effect of the tyrosine kinase inhibitor STI571 in a patient with a metastatic gastrointestinal stromal tumor. N Engl J Med. 2001 Apr 5;344(14):1052-6. doi: 10.1056/NEJM200104053441404. No abstract available. PMID 11287975
- [Background] Camidge DR, Bang YJ, Kwak EL, Iafrate AJ, Varella-Garcia M, Fox SB, Riely GJ, Solomon B, Ou SH, Kim DW, Salgia R, Fidias P, Engelman JA, Gandhi L, Janne PA, Costa DB, Shapiro GI, Lorusso P, Ruffner K, Stephenson P, Tang Y, Wilner K, Clark JW, Shaw AT. Activity and safety of crizotinib in patients with ALK-positive non-small-cell lung cancer: updated results from a phase 1 study. Lancet Oncol. 2012 Oct;13(10):1011-9. doi: 10.1016/S1470-2045(12)70344-3. Epub 2012 Sep 4. PMID 22954507
- [Background] Chow WA, Jiang C, Guan M. Anti-HIV drugs for cancer therapeutics: back to the future? Lancet Oncol. 2009 Jan;10(1):61-71. doi: 10.1016/S1470-2045(08)70334-6. PMID 19111246
- [Background] Kurzrock R, Sherman SI, Ball DW, Forastiere AA, Cohen RB, Mehra R, Pfister DG, Cohen EE, Janisch L, Nauling F, Hong DS, Ng CS, Ye L, Gagel RF, Frye J, Muller T, Ratain MJ, Salgia R. Activity of XL184 (Cabozantinib), an oral tyrosine kinase inhibitor, in patients with medullary thyroid cancer. J Clin Oncol. 2011 Jul 1;29(19):2660-6. doi: 10.1200/JCO.2010.32.4145. Epub 2011 May 23. PMID 21606412